CLINICAL TRIAL: NCT07169357
Title: Efficacy of Hyaluronic Acid Gel and Photobiomodulation Therapy on Wound Healing After Surgical Gingivectomy: A Randomized Controlled Clinical Trial
Brief Title: Testing the Efficacy of Photobiomodulation Therapy and Hyaluronic Acid Gel on Post-surgical Healing After Gingivectomy
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beirut Arab University (Other)
Responsible Party: Principal Investigator, Hanan Rabih Danaf Naim, Principal Investigator, Beirut Arab University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-H-0160-D-M-0692
Record Dates: First submitted 2025-09-05; First posted 2025-09-11 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Gingival Hyperplasia; Gingival Hypertrophy; Gingival Overgrowth; Gingival Enlargement; Photobiomodulation Therapy; Low-level-laser Theraphy
Keywords: LLLT; PBMT; GO; GE
MeSH Terms: conditions — Gingival Hyperplasia; Gingival Hypertrophy; Gingival Overgrowth | interventions — Lasers; Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- test group (Group A) (Active Comparator): Surgical sites after gingivectomy procedures will be irradiated with diode laser (Photobiomodulation therapy) then covered with HA Gel.
  Interventions: Drug: Gengigel; Device: LASER
- test group (Group B) (Active Comparator): Surgical sites will be irradiated with diode laser only
  Interventions: Device: LASER
- control group (group c) (No Intervention): No post-surgical therapy will be performed

INTERVENTIONS:
Drug: Gengigel — The use of Gingigel or 0.2% hyaluronic gel is expected to enhance healing and decrease discomfort in the post-operative period. It exhibits viscoelastic characteristic which serves as osteo-conductive, anti-edematous, antifungal and bacteriostatic effects.
  Other Names: 0.2% hyaluronic acid gel
  Arms: test group (Group A)
Device: LASER — PBMT has markedly been effective in reducing pain, inflammation, edema and postoperative discomfort. It is said to be a natural and effective alternative approach to minimize medicaments prescription such as analgesics, anti-inflammatory or antibiotic drugs. With that said, negative outcomes such as drug side effects, bacterial resistance and post-operative complications can be prevented, thus increasing the success of medical care and assuring a better quality of life
  Other Names: Low-level-laser therapy; low-intensity lasers; non-thermal lasers; cold lasers
  Arms: test group (Group A); test group (Group B)

SUMMARY:
This study consists of random patient selection and allocating them in 3 different groups. After being fit to be included according to the protocol's criteria and signing an informed consent, patients will be distributed after performing a dental surgery known as gingivectomy. Gingivectomy has been classified as the gold standard treatment option for the control of gingival enlargement. Wound recovery after gingivectomy and gingivoplasty occurs by secondary intention healing, thus post-surgical wounds can be strongly associated with discomfort, pain and delayed healing. For that reason, the first group will consist of 13 patients who will be exposed to hyaluronic acid gel or gingigel and photobiomodulation therapy to see if there is significant results in the post-operative healing phase. The second group will also consist of 13 patients who will undergo only photobiomodulation therapy. While the third group will have no clinical supportive care besides follow-up and analgesics upon request.

All the values will be determined by using scores such as Visual analogue scale for pain, Landry's index for healing assessment and oral health quality of life, which consists of 14 questions to asses the enhancement of everyday problems affected by dental situations.

Each case will be followed-up for 3 months post-operative.

DETAILED DESCRIPTION:
The study group consisted of thirty-nine surgical gingivectomy wound sites on patients presenting with gingival hypertrophy on maxillary or mandibular anterior region. Groups will be randomly and equally divided into three groups, Group-A (Test Group 1): Surgical sites after gingivectomy procedures will be irradiated with diode laser (Photobiomodulation therapy) at (940 nm, 0.21 W) with a fiber tip diameter of 400μm for 30 seconds, then covered with HA Gel. Group-B (Test Group 2): Surgical sites will be irradiated with diode laser only at (940 nm, 0.21 W). Group-C (Control Group): No post-surgical therapy will be performed. Wound healing was assessed by implementing Landry, Turnbull and Howley Healing index, while pain perception was objectively evaluated by the patients using the visual analog scale (VAS). To further evaluate the patient's quality of life, Oral Health Impact Profile (OHIP-14) records will be obtained before and after gingivectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patient health ASA I, II
* Average age from 18 to 40 years
* Both genders
* Chronic inflammatory gingival enlargement
* Adequate amount of keratinized tissue.
* Well educated patients as post-operative instructions need to be followed precisely.

Exclusion Criteria:

* Smokers
* Bad oral hygiene
* Allergy to Hyaluronic acid or cosmetic fillers containing H.A
* Any patient under oral contraceptives or immunosuppressive drugs
* Patients undergoing radiotherapy or chemotherapy
* Pregnant or lactating mothers
* Mentally disturbed patients
* Excessive gag reflex
* Patients who refuse to sign informed consent.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2026-02-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Landry's healing index | Wound healing assessed by implementing Landry, Turnbull and Howley Healing index on the 3rd, 7th, 14th, 21st day, 1 month, 2 months and 3 months after the post-surgical procedure.
  to asses the wound healing progress post-surgically in the 3 groups and see how photobiomodulation therapy and the application of hyaluronic acid can enhance the post-operative period.
  Five variables are assessed: tissue color, bleeding on palpation, the presence of granulation tissue, the incision margin and suppuration. It ranges from 1 to 5, with 1 indicating poor healing and 5 indicating excellent healing
Visual analogue scale | Pain perception will be evaluated by using the visual analog scale on the 3rd, 7th, 14th, 21st day and 1 month of periodic follow-up
  to asses the subjected level of pain by the patient throughout the healing process with a minimum score of 0 meaning no pain (best) and a maximum score of 10 meaning severe pain (worse)

SECONDARY OUTCOMES:
Oral health impact profile 14 questions | pre-operative post-operative - on the 7th day - on the 14th day
  to asses the quality of life of patients prior the surgery due to their condition to asses the enhancement of the patient's condition after the surgery and asses how the post-operative interventions bettered their post-operative experience.
  To asses the condition you sum the numerical values of each of the 14 items with a 5-point likert scale 0= never 1= hardly ever 2= ocassionally 3=fairly often 4= very often then you sum the scores of all 14 question to get a total score from 0-56. closer to 56 = greater negative impact of oral health problems on the quality of life closer to 0 =better oral-health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Rania Abdel Fahmy, Phd, Study Director — Beirut Arab University; Nayer Abo Saad, Phd, Study Chair — Beirut Arab University
Locations (1):
- Beirut Arab University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yakout BK, Kamel FR, Khadr MAEA, Heikal LAH, El-Kimary GI. Efficacy of hyaluronic acid gel and photobiomodulation therapy on wound healing after surgical gingivectomy: a randomized controlled clinical trial. BMC Oral Health. 2023 Oct 27;23(1):805. doi: 10.1186/s12903-023-03519-5. PMID 37891549